CLINICAL TRIAL: NCT04169204
Title: Very Old Intensive Care Patients - Perfusion (VIPPER)
Brief Title: Very Old Intensive Care Patients - Perfusion
Acronym: VIPPER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 19-021
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Microcirculation; Intensive Care; Very Old Intensive Care Patients
Keywords: Microcirculation; Intensive Care; Critical care; shock; Very Old Intensive Care Patients; risk stratification; SDF-measurement
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Measurement of microcirculation — As a simple clinical test, every patient will receive the assessment capillary refill time and mottling-score. Additionally, repetitive measurements of lactate will be done. The SDF-camera (MicroVision Medical®, Amsterdam, Netherlands) will measure sublingual microcirculation at different time points (Admission and 24h).

SUMMARY:
Shock is a frequent, etiologically heterogeneous and often lethal clinical condition of intensive care medicine. This is particularly true for very old intensive care patients (VIPs), who are among the fastest-growing subgroups of all intensive care unit (ICU) patients and who suffer from a significantly impaired outcome. In addition to the treatment of the causes of shock, current therapeutic approaches focus on the stabilization of vital parameters, which in general all reflect macrocirculatory measured values such as blood pressure. In contrast, a disturbance of the microcirculation (blood circulation of the smaller blood vessels <100 µm) is only poorly measurable and delayed. The last generation of AVA-Software (MicroVisionMedical) will calculate different parameters about the capillary densitiv and perfusion in a user-independent way. VIPPER investigates whether a non-invasive measurement of microcirculation using the sublingual mucosa in very old intensive care patients in shock leads to faster recognition and specific treatment of organ dysfunctions. Secondly, this study checks whether this measurement predicts outcome.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 80 years
* Acute ICU admission
* Shock at the time point of admission to the ICU or in the first 3 hours defined as Lactate ≥ 2 mmol/l AND need for vasoactive substances to maintain a MAP ≥ 65 mmHg in the presence of adequate volume status

Exclusion Criteria:

* < 80 years
* Inaccessibility for sublingual measurement
* no informed consent

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Very Old Intensive Care Patients with shock
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
bedside measurement of sublingual microcirculation | admission of the intensive care unit
  measurement of sublingual microcirculation by using MicroScan® microscope
bedside measurement of sublingual microcirculation | after 24 hours
  measurement of sublingual microcirculation by using MicroScan® microscope

SECONDARY OUTCOMES:
Mortality | after 30 days, 6 months and 12 months
Length of stay at ICU | tdays from admission of the intensive care unit until discharge
Use of Vasopressors and fluids | days from admission of the intensive care unit until discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bruno RR, Schemmelmann M, Hornemann J, Moecke HME, Demirtas F, Palici L, Marinova R, Kanschik D, Binnebossel S, Spomer A, Guidet B, Leaver S, Flaatten H, Szczeklik W, Mikiewicz M, De Lange DW, Quenard S, Beil M, Kelm M, Jung C. Sublingual microcirculatory assessment on admission independently predicts the outcome of old intensive care patients suffering from shock. Sci Rep. 2024 Oct 27;14(1):25668. doi: 10.1038/s41598-024-77357-y. PMID 39463395